CLINICAL TRIAL: NCT02565589
Title: Hyporesponsiveness of Natural Killer Cells and a Dysfunctional Inflammatory Response in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: NK_ICU_healthy
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICU patient: Critically ill patients who were enrolled less than 24 hours after ICU admission.
- Control: Age-, sex-, and BMI-matched healthy subjects.

SUMMARY:
To investigate natural killer (NK) cell activities, circulating cytokine levels and peripheral blood mononuclear cell (PBMC) cytokine production status in critically ill patients.

DETAILED DESCRIPTION:
Blood samples were collected < 24 hours after admission from 24 intensive care unit (ICU) patients and 24 age-, sex-, and body mass index (BMI)-matched healthy controls. NK cell activities, cytokine concentrations and cytokine production by PBMCs and lipopolysaccharide (LPS)-stimulated PBMCs were measured.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* For healthy controls: nondiabetic and nonobese subjects

Exclusion Criteria:

* For healthy controls: diabetes; history/presence of significant metabolic disease; pregnancy or breast-feeding; acute or chronic infection; liver disease; kidney disease; gastrointestinal disease; subjects taking any drugs or supplements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: From April 2014 to July 2015, 24 critically ill patients were enrolled in this study after admission to the ICU at Yonsei University Severance Hospital. For validation of the experimental findings, age-, sex- and BMI-matched healthy subjects were enrolled as controls among individuals seen at a health evaluation center during the same period.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
NK cell activity | Baseline
  NK cell activity (%)

SECONDARY OUTCOMES:
IL (Interleukin)-12 | Baseline
  IL-12 (pg/mL)
hs-CRP (high-sensitivity C-reactive protein) | Baseline
  hs-CRP (mg/dL)

REFERENCES:
- [Derived] Kim M, Kim M, Jeong H, Chae JS, Kim YS, Lee JG, Cho Y, Lee JH. Hyporesponsiveness of natural killer cells and impaired inflammatory responses in critically ill patients. BMC Immunol. 2017 Dec 8;18(1):48. doi: 10.1186/s12865-017-0231-y. PMID 29221433